CLINICAL TRIAL: NCT03551431
Title: Comparison of Efficacy Between Suggestion Method During Video EEG Recording by Verbal Suggestion in Isolation and Verbal Suggestion Along With Cotton Swab or Tuning Fork for Inducing the Paroxysmal Event in Children Aged 5 to 18 Years With Suspected Psychogenic Nonepileptic Events
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor and Chief, Child Neurology Division, Department of Pediatrics, AIIMS, New Delhi, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Induction
Record Dates: First submitted 2018-05-10; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: EEG, Psychogenic Non Epileptic Events

STUDY DESIGN:
Intervention Model Description: Open labeled, randomized controlled Non-inferiority study with three parallel arms: video EEG with verbal suggestion only, cotton swab with verbal suggestion and tuning fork along with verbal suggestion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video EEG with verbal suggestion (Experimental)
  Interventions: Diagnostic Test: Video EEG with verbal suggestion
- video EEG with verbal suggestion and tuning fork (Experimental)
  Interventions: Diagnostic Test: Video EEG with verbal suggestion
- video EEG with verbal suggestion and cotton swab (Experimental)
  Interventions: Diagnostic Test: Video EEG with verbal suggestion

INTERVENTIONS:
Diagnostic Test: Video EEG with verbal suggestion — Video EEG with verbal suggestion will be done by attaching EEG electrodes to the child along with verbals suggestion in isolation or verbal suggestion and tuning fork, verbal suggestion and cotton swab.

SUMMARY:
In this study we are going to compare efficacy between suggestion method during video EEG recording by verbal suggestion in isolation and verbal suggestion along with cotton swab or tuning fork for inducing the paroxysmal event in children aged 5 to 18 years with suspected psychogenic nonepileptic events. Still there is paucity of data regarding the optimum method for video EEG by suggestion for psychogenic nonepileptic events. We are planning to recruit 25 children aged 5 to 18 years in each of the three arms after taking informed consent from the guardian and then they will be subjected to video EEG by any one of the three suggestion methods.

ELIGIBILITY:
Inclusion Criteria: Children between 5 and 18 years of age with suspected diagnosis of psychogenic nonepileptic events -

Exclusion Criteria: Children with paroxysmal events, who will be later diagnosed as having epilepsy or movement disorder

-

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of children in each group, in whom the paroxysmal event could be reproduced by suggestion | 30 minutes
  Percentage of children in each group, in whom the paroxysmal event could be induced by suggestion

IPD SHARING:
Plan to Share IPD: Undecided